CLINICAL TRIAL: NCT07254520
Title: The Effect of Reiki Therapy on Colic Symptoms and Crying Duration in Infants With Infantile Colic, and on Maternal Fatigue and Quality of Life: A Double-Blind Randomized Controlled Trial
Brief Title: The Effects of Reiki Therapy in Infants With Colic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Duygu Demir, PhD, RN, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: duygudemir Colic
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Reiki; Colic, Infantile
Keywords: Reiki Therapy; Infantile colic; Maternal fatigue; Infant crying; Quality of life
MeSH Terms: conditions — Colic | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The study are conducted based on randomized controlled experimental design with double-blind, pre-test-post-test to determine. The research consists of 2 groups. These groups are Reiki group, control group.
Who Masked: Participant
Masking Description: The research consists of 2 groups. These groups are Reiki group, control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Group (Experimental): Infants in the Reiki group will receive Reiki therapy twice on alternate days, with each session lasting 20-30 minutes, administered by a certified Reiki practitioner following a standardized protocol.
  Interventions: Other: Reiki
- Control Group (No Intervention): Infants in the control group will receive only routine pediatric care and will not receive any Reiki therapy or additional intervention.

INTERVENTIONS:
Other: Reiki — Infants in the Reiki group will receive Reiki therapy twice on alternate days, with each session lasting 20-30 minutes, administered by a certified Reiki practitioner following a standardized protocol.
  Arms: Reiki Group

SUMMARY:
This double-blind, randomized controlled experimental study aims to determine the effect of Reiki therapy administered to infants with infantile colic (aged 3 weeks to 6 months) on infants' colic symptoms and crying duration, as well as on mothers' fatigue levels and quality of life.

The study population consists of infants aged 3 weeks to 6 months who are diagnosed with infantile colic and present to pediatric health and disease outpatient clinics between July 2025 and July 2026. A total of 44 infants meeting the inclusion criteria will be randomly assigned to either the Reiki group (n = 22) or the control group (n = 22).

Data will be collected using the Mother and Infant Descriptive Information Form, the Infantile Colic Scale, the Crying Duration Recording Form, the Visual Analogue Scale for Fatigue (for mothers), and the World Health Organization Quality of Life Scale (WHOQOL) (for mothers).

Reiki therapy will be administered to the intervention group twice on alternate days for 20-30 minutes per session. The control group will not receive any intervention.

DETAILED DESCRIPTION:
The study population consisted of infants aged 3 weeks to 6 months who were diagnosed with infantile colic and met the inclusion criteria, presenting to pediatric health and disease outpatient clinics.

This study was designed as a double-blind, randomized controlled experimental study with a pretest-posttest design to determine the effect of Reiki therapy administered to infants with infantile colic on infants' colic symptoms and crying duration, as well as on mothers' fatigue levels and quality of life.

To ensure homogeneous distribution of the groups, randomization was performed using a computer-based program (http://www.randomization.com

, balanced permutation method). Infants who met the inclusion criteria and whose families agreed to participate were randomly assigned to either the experimental (Reiki) group or the control group according to the randomization list.

The control variables of the study were the infants' demographic characteristics, while the dependent variables were colic pain, crying duration, maternal fatigue level, and maternal quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged between 3 weeks and 6 months.
* Diagnosed with infantile colic by a physician during the study period.
* Birth weight between 2500 and 4000 grams.
* No presence of any chronic disease in the infant.
* Family voluntarily agrees to participate in the study.
* Mother has no visual or hearing impairments.
* Mother is open to communication and cooperation.
* Mother is able to read and understand Turkish.
* Neither the mother nor the infant has received any form of energy therapy (e.g., yoga, Reiki, massage, meditation, or healing touch) within the last five months.

Exclusion Criteria:

* Infants with any acute or chronic illness.
* Infants with congenital anomalies.
* Mothers with diagnosed psychological or mental health disorders.
* Infants diagnosed with lactose intolerance by a physician.
* Infants who have previously been diagnosed with infantile colic and are continuing medical treatment for this condition.

Ages: 3 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Infantile Colic Symptom Score | At baseline and 7th day
  Measured using the Infantile Colic Scale completed by the mother.
Crying Duration of Infants with Infantile Colic | Recorded by the mother over a 7-day period (24 hours per day).
  The mother records the start and end time of each crying episode over a 24-hour period for seven consecutive days to determine the total daily crying duration.
Change in Maternal Fatigue Level | At baseline and 7th day
  Maternal fatigue is assessed using the Visual Analogue Scale for Fatigue (VAS-F), completed by both the mother and an independent nurse. Measurements are taken to evaluate changes in maternal fatigue level.
Change in Maternal Quality of Life | At baseline and 7th day
  Maternal quality of life is assessed using the World Health Organization Quality of Life Assessment (WHOQOL), completed by both the mother and an independent nurse. Measurements are taken to evaluate changes in maternal quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Demir, PhD, Principal Investigator — University of Yalova
Locations (1):
- University of Yalova, Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Den Oudsten BL, Zijlstra WP, De Vries J. The minimal clinical important difference in the World Health Organization Quality of Life instrument--100. Support Care Cancer. 2013 May;21(5):1295-301. doi: 10.1007/s00520-012-1664-8. Epub 2012 Dec 1. PMID 23203652
- [Background] Cirgin Ellett ML, Murphy D, Stroud L, Shelton RA, Sullivan A, Ellett SG, Ellett LD. Development and psychometric testing of the infant colic scale. Gastroenterol Nurs. 2003 May-Jun;26(3):96-103. doi: 10.1097/00001610-200305000-00002. PMID 12811319
- [Background] Pavliuk-Pavliuchenko LL. [An osteotome for the nose]. Stomatologiia (Mosk). 1992 May-Dec;(3-6):84-5. No abstract available. Russian. PMID 1307172
- [Result] Charkhandeh M, Talib MA, Hunt CJ. The clinical effectiveness of cognitive behavior therapy and an alternative medicine approach in reducing symptoms of depression in adolescents. Psychiatry Res. 2016 May 30;239:325-30. doi: 10.1016/j.psychres.2016.03.044. Epub 2016 Mar 30. PMID 27058159
- [Result] Birocco N, Guillame C, Storto S, Ritorto G, Catino C, Gir N, Balestra L, Tealdi G, Orecchia C, Vito GD, Giaretto L, Donadio M, Bertetto O, Schena M, Ciuffreda L. The effects of Reiki therapy on pain and anxiety in patients attending a day oncology and infusion services unit. Am J Hosp Palliat Care. 2012 Jun;29(4):290-4. doi: 10.1177/1049909111420859. Epub 2011 Oct 13. PMID 21998438
- [Result] Wein P, Handler M, Chadda KD. Severe thrombocytopenia as a result of contrast left ventricular angiography. Cathet Cardiovasc Diagn. 1982;8(5):495-9. doi: 10.1002/ccd.1810080511. PMID 6890412
- [Result] Hjern A, Lindblom K, Reuter A, Silfverdal SA. A systematic review of prevention and treatment of infantile colic. Acta Paediatr. 2020 Sep;109(9):1733-1744. doi: 10.1111/apa.15247. Epub 2020 Jun 2. PMID 32150292
- [Result] Icke S, Genc R. Effect of Reflexology on Infantile Colic. J Altern Complement Med. 2018 Jun;24(6):584-588. doi: 10.1089/acm.2017.0315. Epub 2018 Apr 20. PMID 29676928
- [Result] Lecuire J, Dechaume JP, Buffard P, Bochu M. [Meningiomas of the posterior cranial fossa]. Neurochirurgie. 1971 May;17:1-146. No abstract available. French. PMID 4934450
- [Result] Thrane SE, Maurer SH, Ren D, Danford CA, Cohen SM. Reiki Therapy for Symptom Management in Children Receiving Palliative Care: A Pilot Study. Am J Hosp Palliat Care. 2017 May;34(4):373-379. doi: 10.1177/1049909116630973. Epub 2016 Feb 7. PMID 26858170